CLINICAL TRIAL: NCT00761267
Title: A PROSPECTIVE, OPEN-LABEL STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY & EFFICACY OF ANIDULAFUNGIN WHEN USED TO TREAT CHILDREN WITH INVASIVE CANDIDIASIS, INCLUDING CANDIDEMIA
Brief Title: Study To Assess Pharmacokinetics, Safety & Efficacy of Anidulafungin When Treating Children With Invasive Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851008; 2008-004150-32 (EudraCT Number)
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Candidemia
Keywords: Anidulafungin; pediatrics; candidemia; invasive candidiasis; safety
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive | interventions — Anidulafungin; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anidulafungin IV (Experimental): All subjects meeting screening criteria will receive IV anidulafungin.
  Interventions: Drug: Anidulafungin; Drug: Fluconazole

INTERVENTIONS:
Drug: Anidulafungin — Day 1: loading dose of 3 mg/kg (not to exceed 200 mg) Day 2 onwards: maintain a dose of 1.5 mg/kg (not to exceed 100 mg). Minimum total treatment duration is 14 days. Minimum IV anidulafungin treatment duration is 10 days for subjects with microbiologically confirmed ICC and 5 days for subjects at risk of candidiasis; followed by oral fluconazole 6-12 mg/kg/day (not to exceed 800mg/day).
  Maximum treatment duration with anidulafungin is 35 days.
  Other Names: Eraxis
Drug: Fluconazole — Subjects may be switched to oral fluconazole [6-12 mg/kg/day (not to exceed 800mg/day] provided they meet specified criteria. Maximum total treatment duration is 49 days.
  Other Names: Diflucan

SUMMARY:
Prospective, open label study to assess the pharmacokinetics, safety & efficacy of anidulafungin when used to treat children (aged 1 month - <18 years) with invasive candidiasis, including candidemia (ICC).

DETAILED DESCRIPTION:
Prospective, open label study to assess the pharmacokinetics, safety & efficacy of anidulafungin when used to treat children (aged 1 month - < 18 years) with invasive candidiasis, including candidemia (ICC). To participate in the study, at the time of enrollment subjects must (1) have either a confirmed diagnosis of ICC or mycological evidence highly suggestive of Candida sp or (2) in infants 1 month to < 2 years only, be at high risk of candidiasis. All subjects meeting screening criteria receive IV anidulafungin. Subjects will be stratified by age (1 month - < 2 years; 2 years - < 5 years; 5 years - < 18 years). Subjects may be switched to oral fluconazole, provided that the pre-specified criteria are met. Subjects with microbiologically confirmed ICC must have a minimum total treatment duration of 14 days. The maximum allowed treatment duration of anidulafungin is 35 days; the maximum total treatment duration for the study is 49 days. At selected centers, anidulafungin pharmacokinetics will be assessed in the first 6 subjects age 1 month - < 2 years to confirm the recommended dosage regimen. A population PK-PD analysis will be performed in all other enrolled subjects. Subjects will be followed for safety through 6 week FU visit. Efficacy for subjects with confirmed ICC will be assessed at EOIVT, EOT, 2-week FU and 6-week FU visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be either (1) at high risk for candidiasis (1 month - < 2 years ONLY) or (2) have a definitive diagnosis of invasive candidiasis/candidemia (ICC) (All age groups)
* Male and female patients from 1 month to less than 18 years of age.

Exclusion Criteria:

* Any patients with allergy to the drug; and any pregnant female or lactating.
* Failed previous antifungal therapy or expected to live < 3 days.
* Patients with documented or suspected Candida meningitis.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (24):
  - Miller Children's Hospital Bickerstaff Pediatric Family Center, Long Beach, California
  - University of California - Los Angeles, Los Angeles, California
  - University of California - Los Angeles - Ronald Reagan Medical Center, Los Angeles, California
  - University of California - Los Angeles - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Children's Hospital & Research Center Oakland (CHRCO), Oakland, California
  - Children's Hospital of Orange County - Inpatient Pharmacy, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Miami Children's Hospital, Miami, Florida
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland Laboratory University Hospitals Case Medical Center, Cleveland, Ohio
  - Le Bonheur Children's Hospital - 4th Floor, Memphis, Tennessee
  - Le Bonheur Children's Hospital - 7th Floor lab, Memphis, Tennessee
  - LeBonheur Children's Hospital- Central Laboratory, Memphis, Tennessee
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Pediatric Clinical Research Unit University of Tennessee Health Science Center, Memphis, Tennessee
  - Pediatric Clinical Research Unit- 7th Floor Lab, Memphis, Tennessee
  - Pharmacy-University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Tennessee Medical Group Pediatrics, Memphis, Tennessee
  - University of Tennessee Health Science Center, Department of Ophthalmology, Memphis, Tennessee
  - Cook Children's Infectious Diseases Clinic, Fort Worth, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Infectious Diseases Clinic Cook Children's Medical Center, Fort Worth, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Brazil (6):
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba, Paraná
  - Hospital Pequeno Principe, Curitiba, Paraná
  - Hospital Infantil Sabara / Fundacao Jose Luiz Egydio Setubal, São Paulo, São Paulo
  - Instituto PENSI - Pesquisa e Ensino em Saúde Infantil, São Paulo, São Paulo
  - Instituto de Oncologia Pediatrica - Grupo de Apoio ao Adolescente e a Crianca com Cancer, São Paulo, São Paulo
  - Instituto de Oncologia Pediatrica - Grupo de Apoio ao Adolescente e a Crianca com Cancer, São Paulo
- Stollery Children's Hospital - University of Alberta, Edmonton, Alberta, Canada
- Greece (2):
  - Aghia Sophia Childrens Hospital, Athens
  - Hippokration Hospital, Thessaloniki
- Italy (3):
  - Universita degli Studi di Roma La Sapienza, Roma, Province OF ROME
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma, RM
  - Universitario Ospedaliero IRCCS Ospedale Pediatrico Bambino Gesu, Roma, RM
- Russia (2):
  - National Cancer Research Center RAMS n.a. N.N. Blokhin; Laboratory Microbiological Diagnostics, Moscow
  - Fed. Scientific Center for Pediatric Hematology, Oncology and Immunology of Russian Healthcare Org., Moscow
- South Korea (3):
  - Asan Medical Center, Songpa-gu, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Department of Pharmacy, Seoul
- Hospital Vall D'Hebron, Barcelona, Spain
- Taiwan (2):
  - Chang Gung Children's Hospital, Kwei Shan Town, Taoyuan County
  - China Medical University Hospital, Taichung
- Nottingham Children's Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Roilides E, Carlesse F, Tawadrous M, Leister-Tebbe H, Conte U, Raber S, Swanson R, Yan JL, Aram JA, Queiroz-Telles F; Anidulafungin A8851008 Pediatric Study Group. Safety, Efficacy and Pharmacokinetics of Anidulafungin in Patients 1 Month to <2 Years of Age With Invasive Candidiasis, Including Candidemia. Pediatr Infect Dis J. 2020 Apr;39(4):305-309. doi: 10.1097/INF.0000000000002568. PMID 32032174
- [Derived] Roilides E, Carlesse F, Leister-Tebbe H, Conte U, Yan JL, Liu P, Tawadrous M, Aram JA, Queiroz-Telles F; Anidulafungin A8851008 Pediatric Study Group. A Prospective, Open-label Study to Assess the Safety, Tolerability and Efficacy of Anidulafungin in the Treatment of Invasive Candidiasis in Children 2 to <18 Years of Age. Pediatr Infect Dis J. 2019 Mar;38(3):275-279. doi: 10.1097/INF.0000000000002237. PMID 30418357
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851008&StudyName=Study%20To%20Assess%20The%20Safety%2C%20Pharmacokinetics%2C%20And%20Evaluate%20The%20Response%20To%20Anidulafungin%20When%20Treating%20Children%20With%20Invasive%20Candidiasi

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years: Participants received Anidulafungin loading dose of 3 milligrams per kg(mg/kg) intravenously(IV) on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days. After >=10 days treatment, participants with microbiologically confirmed invasive candidiasis/candidemia(ICC) and who fulfilled protocol specified criteria [1)afebrile for >=24 hours, 2)tolerate oral medication, 3)documentation of 2 blood cultures [24 hours apart] negative for Candida, 4)eradication/presumed eradication of Candida from other infection sites,identified at enrollment,5)specific Candida isolate susceptible/presumed susceptible to fluconazole, 6)switched to oral fluconazole if improvement in signs,symptoms of Candida infection] and after >=5 days treatment, participants without microbiologically confirmed ICC,could switch to oral fluconazole(6-12 mg/kg/day,maximum 800mg/day) upto 49 days. First 6 participants received second antifungal agent, if required at Investigator's discretion.
- Anidulafungin: Participants Aged 2 to <5 Years: Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days. After >=10 days treatment, participants with microbiologically confirmed ICC and who fulfilled protocol specified criteria [1)afebrile for >=24 2hours, 2)tolerate oral medication, 3)documentation of 2 blood cultures [24 hours apart] negative for Candida, 4)eradication/presumed eradication of Candida from other infection sites,identified at enrollment,5)specific Candida isolate susceptible/presumed susceptible to fluconazole, 6)switched to oral fluconazole if improvement in signs,symptoms of Candida infection] and after >=5 days treatment, participants without microbiologically confirmed ICC, could switch to oral fluconazole (6-12 mg/kg/day, maximum 800mg/day) for upto 49 days.
- Anidulafungin: Participants Aged 5 to <18 Years: Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days. After >=10 days treatment, participants with microbiologically confirmed ICC and who fulfilled protocol specified criteria ([1)afebrile for >=24 hours, 2)tolerate oral medication, 3)documentation of 2 blood cultures [24 hours apart] negative for Candida, 4)eradication/presumed eradication of Candida from other infection sites,identified at enrollment,5)specific Candida isolate susceptible/presumed susceptible to fluconazole, 6)switched to oral fluconazole if improvement in signs,symptoms of Candida infection]and after >=5 days treatment, participants without microbiologically confirmed ICC, could switch to oral fluconazole (6-12 mg/kg/day, maximum 800mg/day) upto 49 days.
Period: Overall Study
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Started | 20 | 20 | 30
Treated | 19 | 19 | 30
Completed | 18 | 16 | 24
Not Completed | 2 | 4 | 6
Not completed — Death | 1 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Randomized but not treated | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years | Total
Number analyzed (Participants) | 19 | 19 | 30 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.93 (0.52) | 3.09 (0.68) | 10.67 (3.68) | 5.83 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 13 | 30
  Male | 10 | 11 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 19 | 15 | 20 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 6 weeks after end of treatment (EOT) (up to 91 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs. EOT visit defined as last day of study treatment (IV or oral).
Time Frame: Baseline up to 6 weeks after EOT (up to 91 days)
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 19 | 19 | 30
Participants
  AEs | 17 | 19 | 30
  SAEs | 7 | 10 | 13

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hematology parameters: red blood cell count: <0.8*lower limit of normal (LLN); reticulocytes count (absolute or percent): <0.5*LLN or greater than (>) 1.5*upper limit of normal (ULN); Platelets: <0.5*LLN or >1.75*ULN; white blood cell count: <0.6*LLN or >1.5*ULN; neutrophils (absolute or percent): <0.8*LLN or >1.2*ULN; basophils (absolute or percent): >1.2*ULN; lymphocytes (absolute or percent): <0.8*LLN or >1.2*ULN; monocytes (absolute or percent): >1.2*ULN. Serum Chemistry parameters: sodium: <0.95*LLN or >1.05*ULN, potassium, chloride, bicarbonate, calcium: <0.9*LLN or >1.1*ULN; magnesium: >1.1*ULN or <0.9*LLN; BUN (blood urea nitrogen): >1.3* ULN, creatinine: >1.3*ULN; aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase : >3.0*ULN ; total bilirubin: >1.5*ULN; albumin: <0.8*LLN or >1.2*ULN and glucose: <0.6*LLN or >1.5*ULN.EOT visit defined as last day of study treatment (IV or oral).
Time Frame: Baseline up to 6 weeks after EOT (up to 91 days)
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 19 | 19 | 30
Participants | 19 | 18 | 30

3. Secondary Outcome: Number of Participants With Global Response
Description: Global response categorized: success, failure, indeterminate.Success:clinical response(CR) of cure(resolution of sign, symptoms attributed to Candida infection[CI]; no additional systemic/oral antifungal) or improvement (significant but incomplete resolution of signs symptoms of CI; no additional systemic antifungal) and microbiological eradication/presumed eradication(Baseline pathogen not isolated from original site culture/culture data not available for participant with successful outcome).Failure:CR of failure(no significant improvement in signs symptoms/ death due to CI)and/or microbiological failure(persistence/new infection at follow-up/relapse of infection at follow-up). Indeterminate:CR of indeterminate(evaluation not made or failure assessment)and/or microbiological response of indeterminate(Culture data not available for participant with clinical outcome of indeterminate) and neither response was failure.EOT visit:last day of study treatment (IV or oral).
Time Frame: End of intravenous treatment (EOIVT) (maximum of 35 days), EOT (maximum of 49 days), during 2 week follow-up after EOT (up to 63 days) and during 6 week follow-up after EOT (up to 91 days)
Population: The mITT population was defined as all participants who had received at least 1 dose of study drug and who had microbiological confirmation of Candida infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 16 | 18 | 30
Participants
  EOIVT: Success | 11 | 14 | 20
  EOIVT: Failure | 2 | 1 | 3
  EOIVT: Indeterminate | 3 | 3 | 7
  EOIVT: Missing | 0 | 0 | 0
  EOT: Success | 11 | 14 | 21
  EOT: Failure | 2 | 1 | 3
  EOT: Indeterminate | 3 | 3 | 6
  EOT: Missing | 0 | 0 | 0
  2 week follow-up: Success | 11 | 13 | 22
  2 week follow-up: Failure | 2 | 1 | 4
  2 week follow-up: Indeterminate | 3 | 1 | 0
  2 week follow-up: Missing | 0 | 3 | 4
  6 week follow-up: Success | 11 | 12 | 20
  6 week follow-up: Failure | 2 | 2 | 6
  6 week follow-up: Indeterminate | 3 | 2 | 0
  6 week follow-up: Missing | 0 | 2 | 4

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours (AUC24) of Anidulafungin for Pharmacokinetic (PK) Subgroup
Description: Non-compartmental PK analysis was performed on individual plasma anidulafungin concentration-time data collected by serial sampling from participants in the PK sub-study. AUC24 was calculated based on the trapezoidal rule.
Time Frame: Day 2: Just prior to the start of infusion, 2 minutes before the end of infusion, 6, 12 and 24 hours after the start of infusion
Population: PK subgroup population included the first 6 participants aged between 1 month to <2 years.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Anidulafungin PK Subgroup of First 6: 1 Month to <2 Years: First 6 participants received Anidulafungin at loading dose of 3 mg/kg, IV on Day 1, then maintenance dose of 1.5 mg/kg, every 24 hours for minimum of 10 days and maximum of 35 days. After >=10 days of IV treatment, participants with microbiologically confirmed ICC and who fulfilled protocol specified criterion [1) afebrile for >=24 hours, 2) tolerate oral medication, 3)documentation of 2 blood cultures (24 hours apart) negative for Candida species,4) Eradication/presumed eradication of Candida species from any other sites of infection if identified at enrollment, 5) Specific Candida isolate was susceptible/presumed susceptible to fluconazole, 6) switched to oral fluconazole if improvement in signs, symptoms of Candida infection] received oral fluconazole (6 to 12 mg/kg/day, maximum 800 mg/day) up to 49 days. Participants received a second systemic antifungal agent, if required at the Investigator's discretion.
Arm/Group | Anidulafungin PK Subgroup of First 6: 1 Month to <2 Years
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*hr/mL) | 66449.1 (28)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Anidulafungin for Pharmacokinetic (PK) Subgroup
Description: Cmax was obtained directly from the observed concentration data on Day 2.
Time Frame: Day 2: Just prior to the start of infusion, 2 minutes before the end of infusion, 6, 12, and 24 hours after the start of infusion
Population: PK subgroup population included the first 6 participants aged between 1 month to <2 years.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Anidulafungin PK Subgroup of First 6: 1 Month to <2 Years
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL) | 5963.53 (29)

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours (AUC24) of Polysorbate 80 (PS 80) Following Infusion of Anidulafungin for PK Subgroup
Description: Excipient PS 80 is a solubilizing agent contained in the IV formulation of anidulafungin. The lower limit of quantitation (LLOQ) for all the observations of PS 80 was 5.0 microgram per milliliter (mcg/mL). PK time points were assessed on Day 1, Day 3, Day 5, Day 7 and Day 9. Summarized data for all the time points was reported.
Time Frame: Day 1: 0 to 2 hours post dose; Day 3 and Day 9:pre-dose; Day 5: 0 to 3 hours post dose; Day 7: 6 to 12 hours and 24 hours delayed post-dose
Population: The PK subgroup population for PS80 included the last eight participants aged between 1 month to <2 years.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Anidulafungin PK Subgroup of Last Eight: 1 Month to <2 Years: Last eight participants received Anidulafungin loading dose of 3 mg/kg, IV on Day 1, then maintenance dose of 1.5 mg/kg, every 24 hours for minimum of 10 days and maximum of 35 days. After >=10 days of IV treatment, participants with microbiologically confirmed ICC and who fulfilled protocol specified criterion [1) afebrile for >=24 hours, 2) tolerate oral medication, 3)documentation of 2 blood cultures (24 hours apart) negative for Candida species,4) Eradication/presumed eradication of Candida species from any other sites of infection if identified at enrollment, 5) Specific Candida isolate was susceptible/presumed susceptible to fluconazole, 6) switched to oral fluconazole if improvement in signs, symptoms of Candida infection] received oral fluconazole (6 to 12 mg/kg/day, maximum 800 mg/day) up to 49 days. Participants received a second systemic antifungal agent, if required at the Investigator's discretion.
Arm/Group | Anidulafungin PK Subgroup of Last Eight: 1 Month to <2 Years
Number analyzed (Participants) | 8
ng*hr/mL | NA (NA) — Only one value was above LLOQ, hence, AUC24 of polysorbate 80 could not be calculated.

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Polysorbate 80 (PS 80) Following Infusion of Anidulafungin for PK Subgroup
Description: Excipient PS 80 is a solubilizing agent contained in the IV formulation of anidulafungin. The lower limit of quantitation (LLOQ) for all the observations of PS 80 was 5.0 mcg/ml. PK time points were assessed on at Day 1, Day 3, Day 5, Day 7 and Day 9. Summarized data for all the time points was reported.
Time Frame: Day 1: 0 to 2 hours post dose; Day 3 and Day 9:pre-dose; Day 5: 0 to 3 hours post dose; Day 7: 6 to 12 hours delayed post-dose
Population: The PK subgroup population for PS80 included the last eight participants aged between 1 month to <2 years.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Anidulafungin PK Subgroup of Last Eight: 1 Month to <2 Years
Number analyzed (Participants) | 8
ng/mL | NA (NA) — Only one value was above LLOQ, hence, Cmax of polysorbate 80 could not be calculated.

8. Secondary Outcome: Estimated Area Under the Plasma Curve Over a 24-Hour Dosing Interval at Steady State (AUC0-24ss) of Anidulafungin
Description: AUC24 values were calculated using the individual parameter estimates obtained from the final population PK model. PK time points were assessed on Days 1-3, Day 5, Day 7, and Day 9. Data for all time points were included in the model.
Time Frame: Sparse Sampling:Day 1:0-2 hr after end of infusion (EOI); Day3&9:pre-dose;Day 5:0-3hr post EOI; Day 7:6-12hr after EOI.For 1st 6 infants:< 2 years:Day 1:2 minutes before EOI; Day 2:pre infusion, 2 minutes before EOI, 6, 12,24 hours after start of infusion
Population: PK population included all those participants who had 1 or more PK samples available.
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter(mcg*hr/ml)
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 17 | 19 | 30
microgram*hour per milliliter(mcg*hr/ml) | 69.87 (17.65) | 82.81 (31.9) | 86.77 (31.12)

9. Secondary Outcome: Estimated Minimum Plasma Concentration (Cmin) of Anidulafungin
Description: Cmin values were calculated using the individual parameter estimates obtained from the final population PK model. PK time points were assessed on Days 1-3, Day 5, Day 7, and Day 9. Data for all time points were included in the model.
Time Frame: as for outcome 8
Population: PK population included all those participants who had 1 or more PK samples available.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/ml)
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 17 | 19 | 30
microgram per milliliter (mcg/ml) | 1.98 (0.58) | 2.51 (1.11) | 2.52 (0.96)

10. Secondary Outcome: Number of Participants With Greater Than or Equal to 1 Hepatic Adverse Event Categorized on the Basis of Exposure to Anidulafungin (AUC0-24,ss)
Description: The probability of having at least one hepatic adverse event was compared with AUC0-24,ss quantile. Individual parameter estimates from the final PK model were used for estimation of Anidulafungin exposures.
Time Frame: Baseline to End of intravenous treatment (EOIVT) (maximum of 35 days)
Population: Analysis performed on all participants who received at least one dose of the study treatment (Anidulafungin) and had estimable exposure parameters available.
Measure: Count of Participants; unit: Participants
Groups:
- AUC0-24ss (0-61 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss in the range of 0 to 61 mcg*h/ml.
- AUC0-24ss (>61-72 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 61 to 72 mcg*h/ml).
- AUC0-24ss (>72-89 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 72 to 89 mcg*h/ml).
- AUC0-24ss (>89-109 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 89 to 109 mcg*h/ml).
- AUC0-24ss (>109 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 109 mcg*h/ml).
Arm/Group | AUC0-24ss (0-61 mcg*hr/ml) | AUC0-24ss (>61-72 mcg*hr/ml) | AUC0-24ss (>72-89 mcg*hr/ml) | AUC0-24ss (>89-109 mcg*hr/ml) | AUC0-24ss (>109 mcg*hr/ml)
Number analyzed (Participants) | 13 | 18 | 14 | 10 | 11
Participants | 1 | 3 | 5 | 1 | 2

11. Secondary Outcome: Number of Participants With Greater Than or Equal to 1 Gastro-Intestinal (GI) Adverse Event Categorized on the Basis of Exposure to Anidulafungin (AUC0-24,ss)
Description: The probability of having at least one GI adverse event whilst on Anidulafungin treatment was compared with AUC0-24,ss quantile. Individual parameter estimates from the final PK model were used for estimation of Anidulafungin exposures.
Time Frame: Baseline to EOIVT (maximum of 35 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | AUC0-24ss (0-61 mcg*hr/ml) | AUC0-24ss (>61-72 mcg*hr/ml) | AUC0-24ss (>72-89 mcg*hr/ml) | AUC0-24ss (>89-109 mcg*hr/ml) | AUC0-24ss (>109 mcg*hr/ml)
Number analyzed (Participants) | 13 | 18 | 14 | 10 | 11
Participants | 5 | 10 | 6 | 4 | 2

12. Secondary Outcome: Percentage of Participants With Global Response Categorized on the Basis of Exposure to Anidulafungin (AUC0-24,ss)
Description: The probabilities of a global response of success or failure were compared with AUC0-24,ss quantile. Individual parameter estimates from the final PK model were used for estimation of Anidulafungin exposures. For the analysis of this outcome measure, global response was categorized as: success or failure. Success defined as clinical response (CR) of cure (resolution of signs, symptoms attributed to Candida infection [CI]). Failure defined as CR of failure (no significant improvement in signs symptoms/ death due to CI) and/or microbiological failure (persistence/new infection at follow-up/relapse of infection at follow-up).
Time Frame: EOIVT (maximum of 35 days) and EOT (maximum of 49 days)
Population: mITT population: participants who had received at least 1 dose of study drug and who had microbiological confirmation of Candida infection. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and 'Number analyzed' = Participants evaluable for this outcome measure at specified categories.
Measure: Number; unit: percentage of participants
Groups:
- AUC0-24ss (>61-74 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 61 to 74 mcg*h/ml).
- AUC0-24ss (>74-89 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 74 to 89 mcg*h/ml).
- AUC0-24ss (>89-112 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 89 to 112 mcg*h/ml).
- AUC0-24ss (>112 mcg*hr/ml): Participants received Anidulafungin loading dose of 3mg/kg, IV on Day 1 and maintenance dose of 1.5mg/kg, every 24 hours for minimum 10 and maximum 35 days and having AUC0-24ss (more than 112 mcg*h/ml).
Arm/Group | AUC0-24ss (0-61 mcg*hr/ml) | AUC0-24ss (>61-74 mcg*hr/ml) | AUC0-24ss (>74-89 mcg*hr/ml) | AUC0-24ss (>89-112 mcg*hr/ml) | AUC0-24ss (>112 mcg*hr/ml)
Number analyzed (Participants) | 10 | 15 | 9 | 8 | 8
percentage of participants
  EOIVT: Success: number analyzed (Participants) | 10 | 15 | 9 | 8 | 7
  EOIVT: Success | 100 | 93.33 | 77.78 | 87.5 | 85.71
  EOIVT: Failure: number analyzed (Participants) | 10 | 15 | 9 | 8 | 7
  EOIVT: Failure | 0 | 6.67 | 22.22 | 12.5 | 14.29
  EOT: Success | 100 | 93.33 | 77.78 | 87.5 | 87.5
  EOT: Failure | 0 | 6.67 | 22.22 | 12.5 | 12.5

13. Secondary Outcome: Percentage of Participants With Relapsed Response
Description: Relapse was defined as any baseline Candida species isolated following eradication (documented or presumed); or culture data not available for a participant with a clinical response of failure after a previous response of success. Clinical response of failure was defined as no significant improvement in signs and symptoms, or death due to the Candida infection. Participants had received at least 3 doses of study medication to be classified as a failure. Clinical response of success was defined as resolution of sign and symptoms attributed to Candida infection occurred with no additional systemic or oral antifungal treatment required to complete the course of therapy. Eradication or presumed eradication: baseline pathogen not isolated from original site culture(s), or culture data are not available for a participant with successful clinical outcome. End of treatment visit defined as last day of study treatment (IV or oral).
Time Frame: During 2 week follow-up after EOT (up to 63 days) and during 6 week follow-up after EOT (up to 91 days)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 16 | 18 | 30
percentage of participants
  2 week follow-up | 0.0 | 0.0 | 0.0
  6 week follow-up | 0.0 | 5.6 | 6.7

14. Secondary Outcome: Percentage of Participants With New Infection
Description: New infection was defined as a participant presenting with clinical failure with the emergence of new Candida species at the original site of infection or at a distant site of infection. Clinical response of failure was defined as no significant improvement in signs and symptoms, or death due to the Candida infection occurred. Participants had received at least 3 doses of study medication to be classified as a failure. End of treatment visit defined as last day of study treatment (IV or oral).
Time Frame: During 2 week follow-up (up to 63 days) and 6 week follow-up (up to 91 days) after EOT
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 16 | 18 | 30
percentage of participants
  2 week follow-up | 0.0 | 0.0 | 0.0
  6 week follow-up | 0.0 | 0.0 | 0.0

15. Secondary Outcome: All-Cause Mortality - Number of Participants Who Died During Overall Study Treatment Period and Follow-Up Visits
Time Frame: Overall treatment period (up to 49 days); during 2 week follow-up after EOT (up to 63 days) and during 6 week follow-up after EOT (up to 91 days)
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
Number analyzed (Participants) | 19 | 19 | 30
Participants
  overall study treatment period | 0 | 1 | 4
  2 Week Follow-up | 0 | 0 | 1
  6 Week Follow-up | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 6 weeks after end of treatment (up to 91 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety population.
Arm/Group | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years | Anidulafungin: Participants Aged 2 to <5 Years | Anidulafungin: Participants Aged 5 to <18 Years
All-Cause Mortality (participants affected / at risk) | 1/19 | 2/19 | 5/30
Serious Adverse Events (participants affected / at risk) | 7/19 | 10/19 | 13/30
Other Adverse Events (participants affected / at risk) | 17/19 | 17/19 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years (N=19) | Anidulafungin: Participants Aged 2 to <5 Years (N=19) | Anidulafungin: Participants Aged 5 to <18 Years (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Aspiration bronchial (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin:Participants Aged 1 Month to Less Than(<)2 Years (N=19) | Anidulafungin: Participants Aged 2 to <5 Years (N=19) | Anidulafungin: Participants Aged 5 to <18 Years (N=30)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Pupil fixed (Eye disorders) | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Saliva altered (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7 | 5
Catheter site erythema (General disorders) | 0 | 1 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 1
Catheter site rash (General disorders) | 0 | 1 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1
Generalised oedema (General disorders) | 0 | 1 | 1
Hyperpyrexia (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 3 | 6
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 3
Purulent discharge (Infections and infestations) | 0 | 0 | 1
Relapsing fever (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Uterine abscess (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3
Amylase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2
Bacterial test positive (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Enterobacter test positive (Investigations) | 0 | 1 | 0
Klebsiella test positive (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 2
Urine output decreased (Investigations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Areflexia (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 6
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 3 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Henoch-Schonlein purpura nephritis (Renal and urinary disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2
Genital erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haematoma (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 3
Phlebitis (Vascular disorders) | 0 | 0 | 1
Poor venous access (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 2 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Candida test positive (Investigations) | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1
Device dislocation (Product Issues) | 1 | 1 | 0
Device malfunction (Product Issues) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT00761267/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT00761267/SAP_001.pdf